CLINICAL TRIAL: NCT03668899
Title: Assessment of Antimicrobial Efficacy of Nano Chitosan, Chlorhexidine, Chlorhexidine/ Nano Chitosan Combination Versus Sodium Hypochlorite Irrigation in Patients With Necrotic Mandibular Posterior Teeth: A Randomized Clinical Trial
Brief Title: Antimicrobial Efficacy of Four Different Irrigation Protocols
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Maha Nasr, assistant lecturer of Endodontics, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A
Record Dates: First submitted 2018-09-11; First posted 2018-09-13 (Actual); Results first posted 2025-06-29 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Dental Pulp Necrosis
MeSH Terms: conditions — Dental Pulp Necrosis | interventions — Therapeutic Irrigation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Chitosan NPs group (Experimental): irrigation with Chitosan nanoparticles (final flush)
  Interventions: Procedure: irrigation
- Chlorhexidine group (Experimental): irrigation with CHX (final flush)
  Interventions: Procedure: irrigation
- Combination group (Experimental): irrigation with CHX/ nano Chitosan combination (final flush)
  Interventions: Procedure: irrigation
- Hypochlorite group (Active Comparator): irrigation with NaOCL (final flush)
  Interventions: Procedure: irrigation

INTERVENTIONS:
Procedure: irrigation — irrigation of root canals during mechanical preparation for pueposes of cleaning and disinfection

SUMMARY:
proper disinfection of root canal system before obturation is a must for long term success of endodontic treatment, therefore a proper irrigant is mandatory, therefore investigators are studying the antibacterial effects of 4 different irrgating solutions in root canal treatment of patients diagnosed with necrotic pulps in their mandibular posterior teeth. patients will be recruited from outpatient clinic of the endodontic department in cairo university. endodontic treatment will be carried out as usual and samples from the infected root canals will be collected before and after preparation to be cultivated and analyzed at the laboratories of microbiology of faculty of medicine, cairo university

DETAILED DESCRIPTION:
Title:

Assessment of Antimicrobial Efficacy of Nano Chitosan, Chlorhexidine, Chlorhexidine/ Nano Chitosan Combination versus Sodium Hypochlorite Irrigation in Patients with Necrotic Mandibular Posterior Teeth: A Randomized Clinical Trial

Introduction

• Background

Bacteria play a major role in the pathogenesis of apical periodontitis; therefore, success of endodontic treatment is dependent on its complete eradication before obturation1.

It has been established that no instrumentation technique can sufficiently eradicate bacteria from the root canal system without proper irrigation. the success rate of endodontic treatment was claimed to be approximately 10-15% lower for teeth which yield a positive culture before obturation than for teeth which yield a negative culture1.

A verity of irrigating solutions has been introduced and investigated for proper disinfection during endodontic treatment of which sodium hypochlorite (NaOCl) was considered the most popular of all available solutions for its superior antimicrobial effects and tissue dissolving abilities2.

The inability of NaOCl to remove smear layer advocated the use of a chelating agent like EDTA or Citric acid for removal of smear layer after chemo-mechanical preparation3. Yet this wasn't the only downside to the use of NaOCl as the main irrigant, toxicity and irritation to the periapical tissues, burning of the surrounding oral tissues and the weakening effect on dentin flexural strength are also important disadvantages of NaOCl4,5.

Chlorhexidine (CHX), is another popular irrigant which has a broad-spectrum antimicrobial activity plus substantivity, yet it has no tissue dissolving abilities of any kind6. Several studies compared the antimicrobial activity of NaOCl and CHX, some studies showed CHX to be superior to NaOCl7 other studies concluded that it had no added effect to those of NaOCl and that hypochlorite more often achieved negative cultures than CHX8 and several studies proved them both to be similarly effective9.

A wide variety of natural solutions used for irrigation has emerged in order to overcome the downsides of NaOCl including Chitosan nanoparticles. Chitosan nanoparticles are known to have a good antimicrobial activity as well as a chelating effect which will allow for eradication of bacteria and removal of smear layer in the same time10.

• Rationale A. The intervention benefits and databases search results Sodium hypochlorite (NaOCl); the gold standard for irrigation has many disadvantages including irritation of the periapical tissues and burning of surrounding tissues4,5. Therefore, the present study aims to explore new irrigating solutions probably more effective and less irritating to the periapical tissues than NaOCl.

Recent studies have shed the light on a wide range of natural substances like Chitosan, Propolis, and other herbal solutions that are claimed to be as effective against bacteria as NaOCl and less toxic and less irritant4,and also introduced nanoparticles with their known antimicrobial capabilities as endodontic irrigants10,15.

Besides its antimicrobial activity, Chitosan nanoparticles showed promising chelating abilities; Porchena et al suggested that CNPs irrigation was superior to NaOCl in that as well as inhibiting bacterial growth it also can remove the smear layer effectively10.

An in vitro study in 2017 claimed that the combination of 2% Chlorhexidine and 2% Chitosan is as effective as NaOCl against E. Faecalis in biofilms5.

B. The benefits of this study to the population and clinicians It is well established that the most probable cause failure of endodontic treatment is the presence of a persisting infection. Therefore, it is important that chemo-mechanical canal preparation be directed towards complete eradication of all bacteria from the root canal system so that the best possible prognosis can be achieved in endodontic treatment.

Natural alternatives to sodium hypochlorite (NaOCl) can provide as efficient disinfection of the root canal system without the adverse effects of NaOCl on surrounding oral and periapical tissues. This may allow endodontists to perform an efficient and comfortable root canal treatments increasing the patients' confidence and creating a more positive attitude towards the dental profession.

Objective of the present study

The Aim of the current study is to compare the antimicrobial effects of Nano chitosan, Chlorhexidine and Chlorhexidine/ Nano Chitosan combination to sodium hypochlorite in patients with necrotic mandibular posterior teeth

PICO Format

* P: population Patients diagnosed with necrotic mandibular posteriors.
* I: intervention I1: Irrigation with nano chitosan I2: Irrigation with chlorhexidine I3: Irrigation with Chlorhexidine/ nano Chitosan combination
* C: control Irrigation with sodium hypochlorite (NaOCl)
* O: outcome

Primary Outcome

Antibacterial efficacy: will be assessed by counting the number of colony forming units (CFU) after cultivating the collected samples before and after irrigation (S1 and S2) for each patient.

Outcome Tool Unit Time antibacterial efficacy Number of CFUs Numerical data Samples collected before and after preparation and transferred to the laboratory for immediate cultivation.

Secondary outcome Postoperative pain: will be recorded on a visual analogue scale (VAS), pain intensity will be recorded preoperatively and postoperatively after 6, 12, 24,48, 72 hours and 7 days. The VAS consists of a10-cm line anchored by two extremes "No pain" and "pain as bad as could be", patient will be asked to choose the mark that represent their level of pain. Pain level will be assigned to one of 4 categorical scores: 1, None (0); 2, Mild (1-3); 3, Moderate (4-6); 4, Severe (7-10).

Outcome Tool Unit Time Postoperative pain Visual analogue scale VAS Categorial data Immediately after treatment and Up to 7 days after endodontic treatment

Research Question:

In necrotic mandibular posterior teeth, would irrigating the canals using either nano chitosan, chlorhexidine or a combination of nano chitosan and chlorhexidine versus sodium hypochlorite result in better canal disinfection and less postoperative pain?

ELIGIBILITY:
Inclusion Criteria:

1. Patient's age between 22-45 years.
2. Both male and female.
3. Patient who are medically free and with good health
4. Necrotic Mandibular posterior teeth

Exclusion Criteria:

1. Pregnant females.
2. Teeth with vital inflamed pulps, symptomatic periapical abscess and facial cellulitis, periodontally diseased and hopeless teeth.
3. Teeth with previous fillings and/ or previous endodontic treatment

Ages: 22 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2020-01-25 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-08-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maha Nasr, Masters, Principal Investigator — studying for PhD in Cairo University
Locations (1):
- Cairo University, Cairo, Egypt

RESULTS

PARTICIPANT FLOW:
Groups:
- Chitosan NPs Group: irrigation with 3% Chitosan nano particles (final flush)
  irrigation: irrigation of root canals during mechanical preparation for purposes of cleaning and disinfection
- Chlorhexidine Group: irrigation with 2% CHX (final flush)
  irrigation: irrigation of root canals during mechanical preparation for purposes of cleaning and disinfection
- Combination Group: irrigation with 2% CHX/ 3%Chitosan nano particles combination (final flush)
  irrigation: irrigation of root canals during mechanical preparation for purposes of cleaning and disinfection
- Hypochlorite Group: irrigation with 5.25% NaOCL (final flush)
  irrigation: irrigation of root canals during mechanical preparation for purposes of cleaning and disinfection
Period: Overall Study
Arm/Group | Chitosan NPs Group | Chlorhexidine Group | Combination Group | Hypochlorite Group
Started | 15 | 15 | 15 | 15
Completed | 15 | 15 | 15 | 15
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Combination Group: irrigation with 2% CHX/ 3% Chitosan nano particles combination (final flush)
  irrigation: irrigation of root canals during mechanical preparation for purposes of cleaning and disinfection
- Total: Total of all reporting groups
Arm/Group | Chitosan NPs Group | Chlorhexidine Group | Combination Group | Hypochlorite Group | Total
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 60
Age, Continuous [Median (Full Range); unit: years] | 29 [22 to 42] | 31 [24 to 42] | 29 [22 to 41] | 29 [22 to 41] | 30 [22 to 42]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 8 | 8 | 33
  Male | 7 | 6 | 7 | 7 | 27
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Egypt | 15 | 15 | 15 | 15 | 60

OUTCOME MEASURES:

1. Primary Outcome: Number of Colony Forming Units Per Millilitre
Description: activity of the irrigating solution against bacteria in the root canal system, the less the number of colony forming units the better the irrigating solution is
Time Frame: 1 week after culture
Measure: Median (Full Range); unit: CFU/ml
Arm/Group | Chitosan NPs Group | Chlorhexidine Group | Combination Group | Hypochlorite Group
Number analyzed (Participants) | 15 | 15 | 15 | 15
CFU/ml
  preoperative measurements | 80300000 [68900000 to 94100000] | 79900000 [69700000 to 91400000] | 74000000 [51200000 to 96000000] | 73000000 [62700000 to 92400000]
  postoperative measurements | 77000 [52000 to 108000] | 124000 [83000 to 161000] | 88000 [41000 to 104000] | 89000 [51000 to 149000]

2. Secondary Outcome: Numerical Rating Scale
Description: pain incidence and intensity after root canal treatment The NRS consists of an 11 points line anchored by two extremes "No pain" and "pain as bad as could be"
Time Frame: after 6 hours,12 hours, 24 hours, 48 hours, 72 hours and 7 days postoperatively
Measure: Count of Participants; unit: Participants
Arm/Group | Chlorhexidine Group | Chitosan NPs Group | Combination Group | Hypochlorite Group
Number analyzed (Participants) | 15 | 15 | 15 | 15
Participants
  preoperative pain: no pain | 7 | 8 | 6 | 7
  preoperative pain: mild pain | 8 | 7 | 9 | 8
  preoperative pain: moderate pain | 0 | 0 | 0 | 0
  preoperative pain: severe pain | 0 | 0 | 0 | 0
  postoperative pain after 6 hours: no pain | 0 | 0 | 0 | 0
  postoperative pain after 6 hours: mild pain | 0 | 0 | 2 | 2
  postoperative pain after 6 hours: moderate pain | 12 | 10 | 10 | 8
  postoperative pain after 6 hours: severe pain | 3 | 5 | 3 | 5
  postoperative pain after 12 hours: no pain | 0 | 0 | 0 | 0
  postoperative pain after 12 hours: mild pain | 7 | 0 | 8 | 3
  postoperative pain after 12 hours: moderate pain | 7 | 12 | 6 | 11
  postoperative pain after 12 hours: severe pain | 1 | 3 | 1 | 1
  postoperative pain after 24 hours: no pain | 0 | 0 | 0 | 0
  postoperative pain after 24 hours: mild pain | 12 | 11 | 13 | 12
  postoperative pain after 24 hours: moderate pain | 3 | 4 | 2 | 3
  postoperative pain after 24 hours: severe pain | 0 | 0 | 0 | 0
  postoperative pain after 48 hours: no pain | 7 | 7 | 10 | 11
  postoperative pain after 48 hours: mild pain | 8 | 8 | 5 | 4
  postoperative pain after 48 hours: moderate pain | 0 | 0 | 0 | 0
  postoperative pain after 48 hours: severe pain | 0 | 0 | 0 | 0
  postoperative pain after 72 hours: no pain | 13 | 10 | 12 | 11
  postoperative pain after 72 hours: mild pain | 2 | 5 | 3 | 4
  postoperative pain after 72 hours: moderate pain | 0 | 0 | 0 | 0
  postoperative pain after 72 hours: severe pain | 0 | 0 | 0 | 0
  postoperative pain after 7 days: no pain | 13 | 14 | 12 | 13
  postoperative pain after 7 days: mild pain | 2 | 0 | 3 | 2
  postoperative pain after 7 days: moderate pain | 0 | 1 | 0 | 0
  postoperative pain after 7 days: severe pain | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 week
Description: No adverse effects were reported
Arm/Group | Chitosan NPs Group | Chlorhexidine Group | Combination Group | Hypochlorite Group
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15 | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-15): https://cdn.clinicaltrials.gov/large-docs/99/NCT03668899/Prot_SAP_000.pdf